CLINICAL TRIAL: NCT01514435
Title: Clinical Effects of Electroconvulsive Therapy in Severe Depression and Concomitant Changes in Cerebral Glucose Metabolism - an Exploratory Study
Brief Title: Changes in Cerebral Glucose Metabolism After Electroconvulsive Therapy (ECT)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of Graz (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BRECT-2006-PET
Record Dates: First submitted 2012-01-11; First posted 2012-01-23 (Estimated); Last update posted 2012-01-23 (Estimated); Status verified 2012-01

CONDITIONS: Major Depressive Disorder
Keywords: depression; FDG-PET; Electroconvulsive therapy; glucose metabolism
MeSH Terms: conditions — Depressive Disorder, Major; Depression

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- ECT verum group (Experimental): Patients with treatment refractory depression treated with ECT
  Interventions: Device: Electroconvulsive therapy; Device: 18-Fluoro-desoxy-glucose positron emission tomography

INTERVENTIONS:
Device: Electroconvulsive therapy — treatment for major depression
  Other Names: no other names
Device: 18-Fluoro-desoxy-glucose positron emission tomography — intravenous injection of 18-FDG, after 30 min PET-Scan of the brain for aprox. 40 min.
  It´s a neuroimaging technique.
  Other Names: no other names

SUMMARY:
There exist already a few studies that have measured changes of brain metabolism pre and post Electroconvulsive Therapy (ECT) by Positron emission tomography (PET) but these were all performed in a small number of patients and used different methodologies. It is therefore not surprising that these investigations provided inconsistent results, as reviewed previously {{23 Schmidt,E.Z. 2008}}.

In patients with treatment-refractory major depressive episodes, the investigators here therefore probed (a) whether changes in cerebral glucose metabolism measured by PET occur after treatment with ECT and (b) whether these correlate with the clinical amelioration of symptoms. To pursue this goal, the investigators assessed clinical effects, neurocognitive function, and brain metabolism using 18F-Fluoro-deoxyglucose (18F-FDG) PET at baseline and at the end of treatment.

Patients with a treatment refractory depression - defined as absent clinical improvement of depressive symptoms after at least two trials with antidepressants from different pharmacologic classes adequate in dose, duration of at least 6 weeks, and compliance {{30 Berlim,M.T. 2007}} - in whom ECT had been intended on clinical grounds were consecutively asked for participation in this study. Patients had to be between 18 and 80 years old and to be physically healthy.

ELIGIBILITY:
Inclusion Criteria:

* clinical indication for ECT
* treatment refractory depressive episode
* age 18-85 y

Exclusion Criteria:

* addiction as a first diagnosis
* dementia

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2006-05; Primary Completion 2009-05 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
Brain glucose metabolism measured by FDG-PET | one year

CONTACTS AND LOCATIONS:
Overall Officials: Bernd Reininghaus, Principal Investigator — Medical University of Graz
Locations (1):
- Medical University Graz; Department for Psychiatry, Graz, Styria, Austria

REFERENCES:
- [Background] Berlim MT, Turecki G. Definition, assessment, and staging of treatment-resistant refractory major depression: a review of current concepts and methods. Can J Psychiatry. 2007 Jan;52(1):46-54. doi: 10.1177/070674370705200108. PMID 17444078
- [Background] Schmidt EZ, Reininghaus B, Enzinger C, Ebner C, Hofmann P, Kapfhammer HP. Changes in brain metabolism after ECT-positron emission tomography in the assessment of changes in glucose metabolism subsequent to electroconvulsive therapy--lessons, limitations and future applications. J Affect Disord. 2008 Feb;106(1-2):203-8. doi: 10.1016/j.jad.2007.06.009. Epub 2007 Jul 26. PMID 17662472